CLINICAL TRIAL: NCT01819532
Title: Milking the Umbilical Cord Versus Immediate Clamping in Pre-term Infants <33 Weeks: A Randomized Controlled Trial
Brief Title: Milking the Umbilical Cord Versus Immediate Clamping in Pre-term Infants < 33 Weeks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: extremely poor recruitment & since the study was approved, medical practice has evolved to where cord milking is now common practice.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00046760
Record Dates: First submitted 2011-10-06; First posted 2013-03-27 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Prematurity
Keywords: neonate; umbilical cord; cord milking; prematurity
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate umbilical cord clamping (Active Comparator): The umbilical cord will be clamped immediately after delivery.
  Interventions: Procedure: Immediate cord clamping
- Cord milking group (Experimental): The umbilical cord will be "milked" in direction towards neonate 4 times over the course of 10 minutes.
  Interventions: Procedure: Milking group

INTERVENTIONS:
Procedure: Milking group — The umbilical cord will be "milked" toward the neonate four times prior to clamping the umbilical cord.
  Arms: Cord milking group
Procedure: Immediate cord clamping — The umbilical cord will be clamped and cut immediately after delivery of the neonate.
  Arms: Immediate umbilical cord clamping

SUMMARY:
Anemia in preterm neonates is a significant problem encountered frequently in the neonatal intensive care unit. Most preterm neonates born at less than 33 weeks gestation will require at least one blood transfusion during their hospital course and many will require repeated transfusions. Blood transfusions, albeit necessary, carry increased risk of viral infections and transfusion reactions as well as increase the cost of healthcare. The umbilical cord and placenta harbor up to 40% of blood available during fetal life. The current standard of care is immediate umbilical cord clamping. The investigators are performing a randomized controlled trial comparing immediate cord clamping to milking the umbilical cord prior to clamping in neonate born preterm less than 33 weeks gestation. The investigators hypothesize that milking the umbilical cord will demonstrate the same benefits as delayed cord clamping, without delaying neonatal resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates delivered between 24 0/7 and 32 6/7
* Mother carrying a fetus between 24-32 6/7 weeks estimated gestational age
* Written parental consent

Exclusion Criteria:

* Multiple gestation pregnancies (twins or higher order multiples)
* Rh or other antibody sensitization
* Hydrops fetalis
* Known major congenital abnormality
* Suspected abruptio placentae

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin during NICU course | within 24 hours of birth and through NICU stay

SECONDARY OUTCOMES:
1-min Apgar | at 1 minute of life
5 min Apgar | at 5 minutes of life
Blood Sugar upon admission to NICU | within 1 hour of birth
Temperature on admission to NICU | within 1 hour of birth
Cord blood pH | within 1 hour of birth
Blood pressure upon admission to NICU | within 1 hour of birth
Number of volume challenges in first 24 hours of life | at 24 hours of birth
Days requiring ventilation | 2 months
Neonatal death | 6 months
Length of hospital stay | 6 months
Intraventricular hemorrhage | 6 months
Number and volume of blood transfusions | 10 units
duration of phototherapy | 1 month
Maximum serum bilirubin | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Bienstock, MD MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States